CLINICAL TRIAL: NCT07188883
Title: Development of Ege Birth Perception Scale and the Effect of Planned Education on Birth Perception, Birth Fear and Birth Readiness
Brief Title: Development of Birth Perception Scale and Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Selin AHSUN, research assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-7T/9
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Fear of Childbirth
Keywords: birth perception; fear of childbirth; birth readiness; scale development; birth preparation education

STUDY DESIGN:
Intervention Model Description: pretest-posttest, randomized controlled quasi-experimental design intervention research
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): pretest-posttest, randomized controlled quasi-experimental design intervention research
  Interventions: Other: Birth Education
- control group (No Intervention): pretest-posttest, randomized controlled quasi-experimental design intervention research

INTERVENTIONS:
Other: Birth Education — The population consisted of all pregnant women between 24-36 weeks of gestation residing in Izmir province, and the study was completed with a total of 80 pregnant women, 40 pregnant women as intervention and 40 as control in line with the snowball sampling method. Ege Birth Perception Scale, Risk Assessment Form, Individual Introduction Form, Prenatal Self-Assessment Scale, Birth Education Evaluation Form were used to collect the data. Pregnant women who agreed to participate in the study were randomly divided into intervention and control groups; the intervention group received nine hours of online training, while the control group did not receive any intervention.
  Arms: intervention group

SUMMARY:
This study was conducted in two phases. In the first phase, a psychometric instrument was developed and validated to measure women's perceptions of childbirth. The scale demonstrated strong reliability and validity indicators through exploratory and confirmatory factor analyses.

In the second phase, a randomized controlled trial was designed to evaluate the effectiveness of a structured online education program on pregnant women's childbirth-related outcomes. A total of 80 pregnant women were recruited and randomly assigned to either the intervention group (n=40), which received a 9-hour online childbirth education program, or the control group (n=40), which received routine antenatal care.

The primary outcomes were childbirth perception, fear of childbirth, and readiness for birth, assessed at baseline and post-intervention using validated instruments. The results showed that the online education program significantly improved childbirth perception and readiness for birth while reducing fear of childbirth compared to the control group.

This trial provides evidence for the effectiveness of online antenatal education in promoting a positive childbirth experience and may contribute to improving maternal health outcomes in line with international recommendations for respectful maternity care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older
* Gestational age between 20-34 weeks at the time of enrollment
* Ability to read and understand Turkish
* Access to the internet and a device (computer, tablet, or smartphone) to attend online sessions
* Willingness to participate in a 9-hour online childbirth education program
* Provided written informed consent

Exclusion Criteria:

* High-risk pregnancy requiring specialized medical care (e.g., preeclampsia, placenta previa, multiple gestation with complications)
* Known psychiatric disorders that could interfere with participation (e.g., severe anxiety disorder, major depression, psychosis)
* Inability to attend online sessions due to technical or personal limitations
* Previous participation in a structured childbirth education program during the current pregnancy
* Refusal or withdrawal of informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Childbirth Perception Score | Measured by the validated Childbirth Perception Scale at baseline (before intervention) and 4 weeks after the intervention.
Fear of Childbirth Score | Measured by the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) at baseline and 4 weeks after the intervention.
Readiness for Birth Scor | Measured by the Childbirth Readiness Scale at baseline and 4 weeks after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No